CLINICAL TRIAL: NCT06653088
Title: Move Kids-24 h - The Effects of a Physical Education Intervention on Fundamental Movement Skills in Preschoolers
Brief Title: Move Kids-24h Physical Education Program
Acronym: Move Kids-24 h
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Bernardo O'Higgins (Other)
Collaborators: University of Minho (Other); Universidad Mayor (Other); Universidade Lusófona de Humanidades e Tecnologias (Other); Universidade do Porto (Other)
Responsible Party: Principal Investigator, Paz Fernández-Valero, Physical Education Teacher, Universidad Bernardo O'Higgins
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: no 029
Record Dates: First submitted 2024-10-16; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Fundamental Movement Skills; Preschool
Keywords: physical fitness; fundamental movement skills; physical activity; Anthropometrics; Blood pressure
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group with Physical Education program (Experimental): A four-month intervention will be implemented, led by the PE teacher, with three sessions per week. These sessions will last 45 minutes each (Koolwikh et al., 2023), divided into 5 minutes of warm-up, 35 minutes of intervention content, and 5 minutes of return to calm. The program content of the intervention group will contemplate a warm-up with several activities, such as dancing or games. The intervention part will be composed of circuit-based exercises with several stations and games involving locomotion skills, namely run, gallop, slide, skip, jump, hop, etc.; games that integrate manipulative skills, such as throwing, catching, kicking, punting, striking, rolling and bouncing/dribbling; balance games involving swinging, turning, pulling, etc. Games involving perceptual motor skills, such as body schema, laterality, temporality, and spatiality, and games focused on PA. The return to calm will include activities such as yoga, meditation, and flexibility.
  Interventions: Behavioral: Physical Education program
- Control group without programmed PE classes (No Intervention): The control group will continue with their normal activity; however, they will receive the same training after the intervention, so it can also be implemented in their preschools if they wish so (Engel et al., 2022; Santos et al., 2016).

INTERVENTIONS:
Behavioral: Physical Education program — A four-month intervention will be implemented, led by the PE teacher, with three sessions per week. These sessions will last 45 minutes each (Koolwikh et al., 2023), divided into 5 minutes of warm-up, 35 minutes of intervention content, and 5 minutes of return to calm.
  The program content of the intervention group will contemplate a warm-up with several activities, such as dancing or games. The intervention part will be composed of circuit-based exercises with several stations and games involving locomotion skills, namely run, gallop, slide, skip, jump, hop, etc.; games that integrate manipulative skills, such as throwing, catching, kicking, punting, striking, rolling and bouncing/dribbling; balance games involving swinging, turning, pulling, etc. Games involving perceptual motor skills, such as body schema, laterality, temporality, and spatiality, and games focused on PA. The return to calm will include activities such as yoga, meditation, and flexibility.
  Arms: Intervention group with Physical Education program

SUMMARY:
Introduction: The development of fundamental movement skills (FMS) is essential to acquiring the necessary skills that allow children to be competent in several sports, games and dances. Competence is acquired from FMS skills through practice and experiences during childhood. However, evidence from previous studies showed low levels of FMS, given that 4.4% of the preschoolers were delayed in gross motor skills, and 8.8% were at risk of delay.

Aim: To evaluate the effects of a structured physical education (PE) program on preschoolers' FMS, implemented and delivered by PE teachers. Secondary aims are to evaluate the effects of the physical education program on (i) preschoolers' movement behaviors, (ii) physical fitness levels, and (iii) blood pressure.

Methods: Cluster randomized controlled trial study. Sample: 40 preschool children, aged 3 to 4 years old. Primary Outcomes are FMS, assessed with the Test of Gross Motor Development- Third Edition. Secondary outcomes are physical activity (PA), physical fitness, blood pressure and Body Mass Index (BMI).

Expected results: Participation in the PE program will likely have a positive effect on the development of FMS, potentially increasing PA levels and improving physical fitness. It is also expected that FMS show a consistent positive association with BMI and blood pressure levels. The results of this randomized controlled trial (RCT) have the potential to inform future guidelines for PE classes in Chilean preschoolers and strengthen the scientific knowledge on this type of intervention in this population.

DETAILED DESCRIPTION:
Data from children and adolescents has shown that FMS have a significant association and reciprocal longitudinal relationship with PA. Strong evidence to supports a low-to-moderate positive association between FMS and moderate-to-vigorous and vigorous and vigorous PA in preschool-aged children. Conversely, when analyzing results within the 24-hour movement behaviors spectrum, there is evidence that preschoolers who spend more time in sedentary behavior have lower FMS' scores. Short sleep durations can adversely affect the development of FMS. Previous findings also show that proficient FMS may benefit children's physical fitness, specifically cardiorespiratory and musculoskeletal fitness.

FMS' development should begin in the early years; however, data shows that many preschoolers lack adequate FMS proficiency for their age. Additionally, some data show that the Covid-19 worldwide pandemic damaged preschoolers' FMS, together with the motor competence of children aged 6-9 years old, highlighting the need for tailored interventions. Indeed, FMS intervention programs effectively improve FMS, as well as other health-related behaviors and outcomes in preschoolers. Unfortunately, in Chile, many preschools and primary schools do not have structured PE programs, but rather recreation periods in which children participate in free play. However, it has been shown that young children spend only half of their free play time engaged in PA and that PE interventions are an effective mean for developing FMS in preschoolers, but only when implemented by specialized PE teachers. However, in Chile, it is not common to find PE teachers in preschoolers.

Therefore, this research's main aim is to evaluate the effects of a structured PE program on preschoolers' FMS implemented and delivered by PE teachers. The secondary aims are to evaluate the effects of the PE program on (i) preschoolers' movement behaviors, (ii) physical fitness levels, and (iii) blood pressure.

The hypothesis is that a structured physical education program positively modifies fundamental movement skills, movement behaviors, physical fitness levels, and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Preschool children, 3 to 4 years old

Exclusion Criteria:

* Diagnosed physical or mental impairments.

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Fundamental Movement Skills | 2 weeks
  The standardized instrument called the Test of Gross Motor Development (TGMD-3) will be used, which measures 6 locomotor skills (run, gallop, one-legged hop, skip, jump, and slide) and 7 ball skills (two-hand strike, one-hand strike, catch, kick, dribble, overhand throw and underhand throw).

SECONDARY OUTCOMES:
Physical Activity Levels | 5 days
  Accelerometer. The equipment will be placed on the right hip with an adjustable elastic belt. Data will be recorded with an interval of 15 seconds (time) and a frequency of 30 Hz, using Actilife-6 software.
Physical Fitness Levels | 2 weeks
  PREFIT battery encompasses the following tests: handgrip strength for assessing muscular musculoskeletal fitness
Physical Fitness Levels (speed-agility) | 2 weeks
  PREFIT battery encompasses the following tests: The 4x10 m shuttle-run for assessing speed-agility.
Physical Fitness Levels (muscular musculoskeletal fitness) | 2 weeks
  PREFIT battery encompasses the following tests: standing long-jump tests for assessing muscular musculoskeletal fitness.
Body Mass Index (BMI) | 1 day for 10 minutes
  Weight (kg) and height (cm) will be measured, and then the equation kg/m2 will be applied to determine BMI values.
Blood Pressure Levels (systolic and diastolic blood pressure) | 1 day for 15 minutes
  Say here the name of the device. Measured in the right arm, the child will be staying quiet for 3-5 min before measurement, with the back supported and feet uncrossed on the floor.

CONTACTS AND LOCATIONS:
Overall Officials: Paz Fernández-Valero, Principal Investigator — Universidad Bernardo O'Higgins
Locations (1):
- The National Board of Kindergartens, Santiago, Chile

REFERENCES:
- [Background] Santos R, Cliff DP, Howard SJ, Veldman SL, Wright IM, Sousa-Sa E, Pereira JR, Okely AD. "GET-UP" study rationale and protocol: a cluster randomised controlled trial to evaluate the effects of reduced sitting on toddlers' cognitive development. BMC Pediatr. 2016 Nov 9;16(1):182. doi: 10.1186/s12887-016-0723-6. PMID 27829405
- [Result] Garcia-Hermoso A, Alonso-Martinez AM, Ramirez-Velez R, Perez-Sousa MA, Ramirez-Campillo R, Izquierdo M. Association of Physical Education With Improvement of Health-Related Physical Fitness Outcomes and Fundamental Motor Skills Among Youths: A Systematic Review and Meta-analysis. JAMA Pediatr. 2020 Jun 1;174(6):e200223. doi: 10.1001/jamapediatrics.2020.0223. Epub 2020 Jun 1. PMID 32250414
- [Result] Loras H. The Effects of Physical Education on Motor Competence in Children and Adolescents: A Systematic Review and Meta-Analysis. Sports (Basel). 2020 Jun 15;8(6):88. doi: 10.3390/sports8060088. PMID 32549319
- [Result] Hassan MA, Liu W, McDonough DJ, Su X, Gao Z. Comparative Effectiveness of Physical Activity Intervention Programs on Motor Skills in Children and Adolescents: A Systematic Review and Network Meta-Analysis. Int J Environ Res Public Health. 2022 Sep 21;19(19):11914. doi: 10.3390/ijerph191911914. PMID 36231213
- [Result] Engel A, Broderick C, van Doorn N, Hardy L, Ward R, Kwai N, Parmenter B. Effect of a Fundamental Motor Skills Intervention on Fundamental Motor Skill and Physical Activity in a Preschool Setting: A Cluster Randomized Controlled Trial. Pediatr Exerc Sci. 2022 May 1;34(2):57-66. doi: 10.1123/pes.2021-0021. Epub 2021 Oct 25. PMID 34697254